CLINICAL TRIAL: NCT07070791
Title: Investigation of the Effect of Combined Upper Extremity Resistance and Aerobic Exercise Training on Arm Exercise Capacity, Peripheral Muscle Strength and Arm Functionality in Patients With Breast Cancer
Brief Title: Combined Upper Extremity Resistance and Aerobic Exercise Training in Patients With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/5-47
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Upper Extremity; Resistance Exercise; Aerobic Exercise
Keywords: breast cancer; Upper Extremity; resistance exercise training; Aerobic exercise training
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study consisted of two groups: one group performed upper extremity aerobic exercise while the other group performed both upper extremity aerobic exercise and upper extremity progressive resistance training.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Extremity Aerobic Exercise (Active Comparator): Participants will only receive a 12-week upper limb aerobic exercise training program.
  Interventions: Other: Upper Extremity Aerobic Exercise Training
- Upper Extremity Progressive Resistance Training Combined with Aerobic Exercise Training (Experimental): Participants will receive a 12-week upper extremity aerobic exercise training program plus upper extremity progressive resistance exercise training.
  Interventions: Other: Upper Extremity Aerobic Exercise Training; Other: Upper Extremity Progressive Resistance Exercise Training

INTERVENTIONS:
Other: Upper Extremity Aerobic Exercise Training — 12 weeks of upper extremity aerobic exercise training, 3 sessions per week, 25 minutes per session.
Other: Upper Extremity Progressive Resistance Exercise Training — Upper extremity progressive resistance training was gradually increased over 12 weeks using elastic resistance bands.
  Arms: Upper Extremity Progressive Resistance Training Combined with Aerobic Exercise Training

SUMMARY:
According to updated data from the International Agency for Research on Cancer (IARC) for 2022, breast cancer in women is responsible for one in four cancer cases and one in six cancer deaths worldwide and is the second leading cause of global cancer incidence, accounting for 11.6% of all cancer cases, and the fourth leading cause of cancer deaths worldwide, accounting for 6.9% of all cancer deaths. During or after breast cancer treatments, there is exposure to a variety of direct (local/regional treatment, systemic treatment and supportive care) and indirect factors (modifiable and non-modifiable risk factors) that may have adverse effects on treatment-related haematological, cardiovascular, pulmonary and musculoskeletal components. Upper limb dysfunction and lymphoedema have been reported to be two of the most common side effects affecting the quality of life of breast cancer patients after breast cancer treatments. The elastic resistance band, which is widely used in strength training, has the advantage of being applied to various classes because it provides resistance angles in various postures and has a low risk of injury. However, few studies have been conducted on elastic resistance band application in patients with breast cancer. At the same time, evidence on the effectiveness of upper extremity aerobic exercise training in patients with breast cancer is limited. Therefore, this study aimed to investigate the effects of upper extremity aerobic exercise training combined with progressive resistance training and upper extremity aerobic exercise training alone on upper extremity exercise capacity, upper extremity functionality, sarcopenia, frailty, quality of life and lymphedema in patients with breast cancer.

DETAILED DESCRIPTION:
According to updated data from the International Agency for Research on Cancer (IARC) for 2022, breast cancer in women is responsible for one in every four cancer cases and one in every six cancer deaths worldwide and is the second leading cause of global cancer incidence, accounting for 11.6% of all cancer cases, and the fourth leading cause of death from cancer worldwide, accounting for 6.9% of all cancer deaths. The prognosis of breast cancer has improved significantly with comprehensive screening programmes, early diagnosis and innovative systematic treatments, with a 5-year survival rate of 90% and a 10-year survival rate of approximately 80%. On the other hand, with increasing survival rates, various strategies are needed for the management of short- and long-term sequelae related to breast cancer treatments, especially considering quality of life. During or after breast cancer treatments, patients are exposed to various direct (local/regional treatment, systemic treatment and supportive care) and indirect factors (modifiable and non-modifiable risk factors) that may have adverse effects on haematological, cardiovascular, pulmonary and musculoskeletal components. Upper limb dysfunction and lymphoedema have been reported to be two of the most common side effects affecting the quality of life of breast cancer patients after breast cancer treatments. Up to 70% of breast cancer patients experience pain, discomfort and/or reduced physical function in the affected shoulder, arm and hand, depending on the type of surgery, rehabilitation programmes or assessment tools and other factors. The percentage of women experiencing lymphoedema after breast cancer surgery is very heterogeneous and varies between studies from 4% to over 60%. As a result of upper extremity dysfunction, decreased ability of individuals to perform activities of daily living is frequently observed. This is a major concern in terms of clinical and public health. In addition, the increase in arm volume and lymphoedema represent a significant threat to life. The American Cancer Society and the National Cancer Institute recommend exercise led by an expert as a safe and feasible method to reduce the risk of developing lymphoedema. Furthermore, many studies have observed that resistance training and concurrent training are beneficial in preventing short- and long-term upper extremity disorders. Resistance training and other forms of physical activity are among the most effective treatments to regain shoulder joint mobility, reduce pain and discomfort, and improve quality of life in breast cancer patients. In addition, some studies suggest that resistance exercise may reduce lymphoedema. However, there is still a lack of information for patients due to medical recommendations to restrict the affected arm and a lack of implementation of these recommendations in clinical practice, leading to greater fear of using the affected arm, lower physical activity, lower muscle strength and greater perceived weakness.

The elastic resistance band, which is widely used in strength training, has the advantage of being applied to various classes because it provides resistance angles in various postures and has a low risk of injury. However, few studies have been conducted on elastic resistance band application in patients with breast cancer. At the same time, evidence on the effectiveness of upper extremity aerobic exercise training in patients with breast cancer is limited. Therefore, this study aimed to investigate the effects of upper extremity aerobic exercise training combined with progressive resistance training and upper extremity aerobic exercise training alone on upper extremity exercise capacity, upper extremity functionality, sarcopenia, frailty, quality of life and lymphedema in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18-80 years old,
* Volunteering to participate in the research,
* At least 15 months after breast cancer surgery,
* No problems in reading and/or understanding the scales and being able to co-operate with the tests.
* Physically inactive (60 minutes of structured exercise per week <).

Exclusion Criteria:

* Presence of active infection,
* Presence of bilateral breast cancer,
* History of surgical, neurological or orthopaedic problems that may affect upper extremity functionality other than breast cancer surgery,
* Having a neurological disease or other clinical diagnosis that may affect cognitive status,
* Musculoskeletal and neurological disease that may affect exercise performance, symptomatic heart disease, previous lung surgery and malignant disease.
* Presence of unstable hypertension or diabetes mellitus.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
6 minute Pegboard and Ring Test - 6PBRT | One Year
  Total number of rings inserted in six minutes
Maximal Arm Exercise Capacity | One Year
  VO2peak requirement during arm ergometry will be estimated using MET levels calculated at each power output based on gender at various body weights and will be displayed in ml/kg/min (1 MET = 3.5 ml/kg/min)

SECONDARY OUTCOMES:
Evaluation of Quality of Life | One Year
  European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) All scores were linearly transformed to a 0 to 100 scale. A high or healthy level of functioning is represented by a high functional score
Peripheral Muscle Strength | One Year
  Hand grip strength by hand dynamometer
Anthropometric Measurements | One Year
  Arm Circumference
Comorbidity Assessment | One Year
  The Charlson Comorbidity Index According to this index developed by the Institute of Medicine, comorbid diseases are assessed according to their severity. is scored. Comorbidities are scored from mild disease state to severe disease state. are given a score of 1, 2, 3, 4, respectively, and the score obtained by summing the scores of comorbid diseases The severity of comorbidity is also calculated according to the weighted score. One point for every ten years over the age of forty (50-59: 1 point, 60-69: 2 points, etc.)
Peripheral muscle strength assessment | One Year
  Peripheral muscle strength (knee extensors, shoulder abductors and hand grip strength) will be measured using a handheld digital dynamometer
Evaluation of Upper Extremity Functionality | One Year
  Questionnaire Disability of Arm, Shoulder and Hand (Q-DASH) Each item is scored on a 5-point Likert scale (1-5).The maximum score is 100 points. Score increase shows an increase in disability.
Assessment of Sarcopenia | One Year
  According to EWGSOP2, probable sarcopenia is defined by the first criterion and confirmed sarcopenia by the first and second criteria. Severe sarcopenia is considered if all three criteria are present.
Assessment of Frailty Status | One Year
  Those who do not fulfil any of the criteria are defined as non-fragile group and those who fulfil 1 or 2 of the criteria are defined as pre-fragile group.
Lymphoedema Evaluation | One Year
  Using circumference measurements starting from the wrist, the volume of the upper extremity was calculated by using an excel programme (Calculator: John Chambers) which calculates the volume by taking the sum of the volumes of truncated cones standing on top of each other. Lymphedema was considered positive in patients with a volume difference of more than 200 ml between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Melda Saglam, PhD, Study Chair — Hacettepe University; Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hcettepe University, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No